CLINICAL TRIAL: NCT06004167
Title: 5-5-5 Adaptive Bridging Radiation Therapy (ABRT) for Relapsed/Refractory B-cell Lymphoma Prior to CAR T-cell Therapy
Brief Title: Adaptive Bridging RT in R/R B-cell Lymphoma (Pre-CAR T)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Chirayu Patel, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-364
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma, B-Cell; Relapsed Cancer; Refractory Lymphoma; Diffuse Large B Cell Lymphoma; Mediastinal Large B-cell Lymphoma; High-grade B-cell Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma
Keywords: Relapsed/Refractory B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence; Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 5-5-5 Adaptive Bridging Radiation Therapy (ABRT) (Experimental): 5 Gy of adaptive radiation delivered every 5 business days (1 week apart) for up to 5 weeks prior to CAR T-cell therapy infusion
  Interventions: Radiation: Adaptive Bridging Radiation Therapy (ABRT)

INTERVENTIONS:
Radiation: Adaptive Bridging Radiation Therapy (ABRT) — Radiation Therapy

SUMMARY:
Participants are invited to take part in this research study because they have relapsed (cancer has come back) or refractory (cancer has not responded to treatment) B-cell Lymphoma and will be undergoing CAR T-cell Therapy.

This research is being done to see if a new radiation therapy administration schedule will positively impact the logistics, time, cost, and side effects of radiation therapy.

In this research study, participants will receive radiation therapy once weekly for 5 weeks. This is a novel administration schedule and we're looking to see how this schedule impacts side effects participants may experience, the time spent receiving radiation therapy, how much radiation therapy participants can receive, and how effective this new schedule is.

DETAILED DESCRIPTION:
This is a feasibility/pilot study of 5 Gy adaptive radiation administered every 5 business days (1 week apart) for 5 weeks prior to standard of care CAR T-cell therapy infusion. Approximately 10 participants with Relapsed/Refractory B-cell Lymphoma will take part in this research study. The primary objective is to assess the feasibility of once weekly radiation therapy for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed or refractory B-cell lymphoma (including, but not limited to diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B-cell lymphoma, high grade B-cell lymphoma, DLBCL arising from follicular lymphoma, follicular, and mantle cell lymphoma)
* Being planned to undergo CAR T-cell therapy (patients can be enrolled prior to apheresis)
* At least 1 measurable lesion according to the Lugano criteria35. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy. Re-irradiation is allowed for these patients. More than 1 lesion can be targeted as per radiation oncologist discretion. If disease is palpable, physical examination alone may be sufficient measurement for disease if a recent PET/CT or CT is not available as a radiologic measurement of the disease can be obtained during CT simulation.
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 3.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any medical condition likely to interfere with assessment of safety or efficacy of RT.
* CNS-only disease as the site for bridging radiation therapy (which cannot be reliably evaluated on CT). Patients with CNS disease with extra-axial involvement that can be evaluated on CT remain eligible.
* Patient likely unable to lay supine for 45 minutes
* Women of child-bearing potential who are pregnant because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant. Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential
* In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-14 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Feasibility: Percent of patients able to undergo ABRT | 20 months
  Feasibility is being measured based on the percentage of patients being able to undergo ABRT

SECONDARY OUTCOMES:
Adverse Events | 20 months
  Adverse events will be classified and graded according to the CTCAE v.5.0.
Objective Response Rate (ORR) | 15 months
  ORR is being measured using the day 30 and day 90 PET scans and assessed by Lugano lymphoma response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Chirayu Patel, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Ababneh HS, Ng AK, Wan J, Walburn T, Zhu L, Bobic M, Johnson PC, Bredtfeld J, Leeman J, Soumerai J, Abramson JS, Barnes J, Takvorian R, Frigault MJ, Pursley J, Patel CG. 5-5-5 ABRT (Dose of 5 Gy per Fraction for up to 5 Fractions Over 5 Weeks Adaptive Bridging Radiation Therapy)-Artificial Intelligence Enters the CAR (-T) (Chimeric Antigen Receptor-T) in Relapsed/Refractory Large B Cell Lymphoma. Int J Radiat Oncol Biol Phys. 2025 Jul 15;122(4):936-948. doi: 10.1016/j.ijrobp.2025.03.023. Epub 2025 Apr 3. PMID 40178467